CLINICAL TRIAL: NCT03324022
Title: Observing the Relationship of Fibroblast Growth Factor and Fibroblast in Thyroid Eye Disease
Acronym: TED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412026RINB
Record Dates: First submitted 2017-10-16; First posted 2017-10-27 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Graves Ophthalmopathy
Keywords: Fibroblast growth factors; Fibroblast growth factors receptors; Thyroid orbitopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Graves' orbitopathy (GO) affects about 50% of patients with Graves' disease (GD), and some cannot be cured by current treatments. Orbital fibroblasts involves in the pathogenesis of GO by producing glycosaminoglycans and inflammatory cytokines. Since fibroblast growth factors (FGFs) binding to FGF receptors (FGFRs) can induce proliferation and differentiation of fibroblasts, investigators would like to measure the expression of FGFs and FGFRs in GO patients to see if inhibition of FGF-FGFR pathway has potential in treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as thyroid eye disease
* suggested to accept orbital decompression

Exclusion Criteria:

* age below 20 or above 80
* pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid eye disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-12-25 (Actual); Primary Completion 2017-12-25 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of selected growth factors | 1 year
  Investigators would like to measure fibroblast growth factors concentration (ug/mL) by ELISA according to the manufacturers' instruction

SECONDARY OUTCOMES:
RNA expression level of selected growth factor receptors | 1 year
  Investigators would like to measure growth factor receptors expression level comparing to house-keeping gene using real-time PCR
RNA expression level of selected growth factor receptors | 1 year
  Investigators would like to measure adipogenesis-related genes expression level comparing to house-keeping gene using real-time PCR

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Derived] Shih SR, Liao SL, Shih CW, Wei YH, Lu TX, Chou CH, Yen EY, Chang YC, Lin CC, Chi YC, Yang WS, Tsai FC. Fibroblast Growth Factor Receptor Inhibitors Reduce Adipogenesis of Orbital Fibroblasts and Enhance Myofibroblastic Differentiation in Graves' Orbitopathy. Ocul Immunol Inflamm. 2021 Jan 2;29(1):193-202. doi: 10.1080/09273948.2019.1672196. Epub 2019 Oct 28. PMID 31657648